CLINICAL TRIAL: NCT05188495
Title: Phase II Study of Trastuzumab(Henlius®) Combined With Pertuzumab(Perjeta®) and Chemotherapy in Chinese Patients With Human Epidermal Growth Factor Receptor 2-Positive Metastatic Breast Cancer Previously Treated With Trastuzumab
Brief Title: Trastuzumab(Henlius®) Combined With Pertuzumab(Perjeta®) and Chemotherapy in Chinese Patients With Her2-Positive Metastatic Breast Cancer Previously Treated With Trastuzumab
Acronym: HELP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Li Huiping, Director of Breast oncology department, Peking University Cancer Hospital & Institute
Other Study IDs: 2020KT151
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: HER2-positive Metastatic Breast Cancer; Previously Treated With Trastuzumab; Trastuzumab Combined With Pertuzumab and Chemotherapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: trastuzumab(Henlius®) combined with Pertuzumab(Perjeta®) and Chemotherapy — trastuzumab(Henlius®) combined with Pertuzumab(Perjeta®) and Chemotherapy； TPC:treatment of physician's choice,include taxanes，Gemcitabine, capecitabine, vinorelbine

SUMMARY:
Currently, data of the efficacy of trastuzumab plus pertuzumab and chemotherapy is limited in the HER2 positive metastatic breast cancer patients previously treated with trastuzumab during (neo)adjuvant and metastatic setting, and results are not consistent.The main purpose of this study is to evaluate the 6-month progression free survival(PFS) of trastuzumab(Henlius®) combined with Pertuzumab(Perjeta®) and Chemotherapy as first to third line therapy in Chinese patients with HER2 positive metastatic breast cancer who received trastuzumab previously.Primary Endpoint is 6-month Progression-free survival (PFS);Secondary Endpoint(s) include Progression-free survival (PFS) Overall Survival (OS);Objective Response Rate(ORR);

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

  1. Adults ≥18 years old
  2. Histologically confirmed invasive BC: incurable, immunohistochemistry (IHC) 3 + or fish confirmed gene amplification: HER2 / CEP 17 ratio ≥ 2, and either of the two analysis results is positive.
  3. Patients with metastatic breast cancer previously treated with trastuzumab 1) the number of lines receiving anti-HER2 treatment for metastatic diseases was 0-2 2) If the number of lines previously receiving anti-HER2 treatment for metastatic diseases is 0, it is required that the last time of preoperative( neoadjuvant) and / or postoperative (adjuvant) trastuzumab is more than 6 months before recurrence and metastasis.
  4. Measurable disease as defined per RECIST v.1.1. Patients with only central nervous system diseases are not suitable for inclusion.
  5. Left ventricular ejection fraction (LVEF) ≥ 50%, determined by echocardiography.
  6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
  7. Adequate organ and bone marrow function defined as follows,Confirmed by the following laboratory examination results within 7 days before randomization：

     * (1) Absolute Neutrophil Count (ANC) ≥1,500/mm3 (1.5 x 109 /L);
     * (2)Platelets ≥100,000/mm3 (100 x 109 /L);
     * (3) Hemoglobin ≥9 g/dL (90 g/L);（patients are allowed to reach these levels through blood transfusion or drug treatment）
     * (4)Albumin ≥ 2.5 g / dl
     * (5)Serum creatinine ≤1.5 x Upper Limit of Normal (ULN)
     * (6)Total serum bilirubin ≤1.5 x ULN (≤3.0 x ULN if Gilbert's disease);
     * (7) AST and/or ALT ≤3 x ULN (≤5.0 x ULN if liver metastases present);
     * (8) INR and APTT < 1.5 ´ upper normal limit (ULN) (unless receiving anticoagulant therapy);
  8. Women with fertility: agree to abstinence (no heterosexual intercourse) or use non hormonal contraceptive methods with an annual failure rate of less than 1% during treatment and at least 7 months after the last administration of the test drug.

     If a female patient is in the late menopause, has not yet reached the postmenopausal state (continuous non menstruation time ≥ 12 months, and there is no other confirmed reason except menopause), and has not received sterilization surgery (removal of ovary and / or uterus), the patient is considered to be fertile.

     Examples of non hormonal contraceptive methods with an annual failure rate of < 1% include bilateral tubal ligation, male contraception and copper ring IUD.

     Barrier contraception must be supplemented by spermicide. Alternatively, use two methods at the same time (e.g. two barrier contraceptives, such as condoms and uterine caps) to achieve an annual failure rate of < 1%.
  9. Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Patients presenting with any of the following will not be included in the study:

  1. History of receivingpatuzumab in the treatment of metastatic diseases (if used during adjuvant or neoadjuvant, the time from the last medication to recurrence and metastasis should be more than 12 months)
  2. History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage 1 uterine cancer, synchronous or previously diagnosed HER2-positive BC, or cancers with a similar curative outcome as those mentioned above
  3. History of receiving chemotherapy or trastuzumab within 21 days before randomization (7 days in the case of weekly regimen)
  4. History of radiation therapy within 14 days before randomization
  5. Patients must recover from acute toxicity caused by previous treatment (to ≤ grade 1) before randomization.
  6. Untreated symptomatic progressive brain metastases occurred within 30 days before randomization.
  7. The cumulative dose of exposure to the following anthracyclines is detailed as follows:

     Doxorubicin > 500 mg/m2 Epirubucin > 720 mg/m2 Mitoxantrone > 120 mg/m2 If other anthracyclines or several anthracyclines are used, the cumulative dose must be less than the equivalent dose of 500 mg / m2 adriamycin.
  8. Current unstable ventricular arrhythmia requiring treatment.
  9. History of symptomatic congestive heart failure（CHF， [NYHA]II-IV级）。
  10. History of myocardial infarction or unstable angina within 6 months of enrollment
  11. History of a decrease in LVEF to < 50% or symptomatic CHF with previous trastuzumab treatment
  12. Severe dyspnea at rest due to complications of advanced malignancy or requiring current continuous oxygen therapy
  13. Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease)
  14. Pregnancy or lactation
  15. Currently known active infection with HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV).

For patients who are known carriers, active HBV infection must be ruled out. Active HBV infection is defined on the basis of results of three tests: positive HBsAg, detectable HBV DNA, and ALT > ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients with HER2 positive metastatic breast cancer who received trastuzumab previously in first to third line setting
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-12-10 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
6-month Progression-free survival (PFS) rate | from the day treatment started to 6 months
  the proportion of patients who were progression free at 6 months or later. were progression free at 6 months or later.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruyan Zhang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang R, Liu X, Song G, Zhang Y, Li H. Trastuzumab Biosimilar (HLX02), Pertuzumab Plus Chemotherapy in Patients with HER2-Positive Metastatic Breast Cancer after Progression of Trastuzumab: A Prospective, Phase II Study. Cancer Res Treat. 2024 Jul;56(3):795-801. doi: 10.4143/crt.2023.1151. Epub 2023 Dec 20. PMID 38147816